CLINICAL TRIAL: NCT04359693
Title: Impact of SARS-CoV-2 Infection on the Incidence of Ventilator-acquired Infections
Brief Title: Impact of COVID-19 Infection on the Incidence of Ventilator-acquired Infections
Acronym: COVAPID
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2020_27; 2020-A00995-34 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: SARS-CoV 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- SARS-CoV2 group: Patients receiving invasive mechanical ventilation for more than 48h with SARS-CoV-2 infection
- Flu group: Patients receiving invasive mechanical ventilation for more than 48h with influenza infection
- No viral infection group: Patients receiving invasive mechanical ventilation for more than 48h with no viral infection at ICU admission

SUMMARY:
Observational cohort study aiming at comparing the incidence of ventilator-associated lower respiratory tract infections between COVID-19 patients and two control groups: one with influenza pneumonia and the other with no viral pneumonia.

DETAILED DESCRIPTION:
COVAPID is a multicenter cohort study with two retrospective control groups. No intervention will be performed in included patients, only patient characteristics and data on VA-LRTI will be collected.

Patients with confirmed SARS-CoV-2 community-acquired pneumonia, admitted to the participating ICUs from the start of COVID epidemic will be eligible for this study. Those admitted before the beginning of this study will be included retrospectively, and those admitted after the beginning of the study will be included prospectively. 10-20 patients per center will be included in this group. SARSCoV2 infection will be confirmed by a nasopharyngeal PCR or respiratory secretions (tracheal aspirate or bronchoalveolar lavage) PCR. Two retrospective groups will be constituted in order to give some insight of potential impact of SARS-CoV2 infection on the incidence of VALRTI :1) Influenza group : patients with influenza (A or B) community-acquired pneumonia. All patients with influenza community acquired pneumonia and admitted in the same ICU will be eligible in this group.

The number of patients included in this group per center will be similar as that of patients included in the SARS-CoV-2 pneumonia group (10-20 patients). These consecutive patients will by identified using the files of Virology Lab. The first included patient will be the last of the current influenza season (2019-2020), and others will be taken consecutively back to 2019 of 2018 if necessary. PCR (nasopharyngeal or respiratory secretions) confirmation of influenza (A ou B) is required for patients in this group. 2) No viral infection group: patients with no viral community acquired pneumonia. All patients receiving invasive mechanical ventilation for more than 48h before COVID epidemic, for any reason other than viral pneumonia are eligible for this group. The number of included patients in this group will be similar as that of patients included in the SARS-CoV-2 group in the same center (10-20 patients) These consecutive patients will be included starting at the end of January 2020 and going back to 2019 if necessary. VAT and VAP are defined using clinical, radiological and quantitative microbiological criteria.

ELIGIBILITY:
Inclusion Criteria:

For all three groups:

* Major patient
* In patients in ICU
* Patients intubated and mechanically ventilated for more than 48 hours.

For the SARS-CoV2 group: community-acquired SARS-CoV2 pneumonia For the influenza group: community-acquired influenza pneumonia For the "No Viral Infection" group: no viral pneumonia on admission.

Exclusion Criteria:

* Refusal to participate
* Lack of social security coverage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients suspected of pulmonary infection and admitted in ICU
Sampling Method: Non-Probability Sample
Enrollment: 1576 (Actual)
Dates: Start 2020-04-22 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of ventilator-associated lower respiratory tract infection | from day 3 of mechanical ventilation to extubation or day 28 post-intubation.
  the incidence of ventilator associated pneumonia and ventilator associated tracheobronchitis

SECONDARY OUTCOMES:
Cumulative incidence of ventilator-associated tracheobronchitis | from day 3 of mechanical ventilation to extubation or day 28 post intubation
  incidence of ventilator-associated tracheobronchitis
Cumulative incidence of ventilator-associated pneumonia | from Day 3 of mechanical ventilation to extubation or day 28 post intubation.
  incidence of ventilator-associated pneumonia
the cumulative incidence of ICU acquired bacteremia diagnosed | from ICU admission to extubation or Day 28.
  incidence of ICU-acquired bacteremia
ICU mortality | at day 28
  death in the ICU
Mortality | at day 28
  death
the duration of mechanical ventilation | from the start of mechanical ventilation to extubation or day 28 post intubation
  number of days Under mechanical ventilation
Length of stay in Intensive Care Unit | from admission to ICU until extubation or Day 28
  number of days in the ICU

CONTACTS AND LOCATIONS:
Overall Officials: Saad Nseir, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Roger Salengro, ICU, CHU Lille, Lille, France

REFERENCES:
- [Derived] Kreitmann L, Bayon C, Martin-Loeches I, Povoa P, Salluh J, Rouze A, Moreau AS, Duhamel A, Labreuche J, Nseir S; Type of iMmunosuppression and the Incidence, Microbiology, and OutcomeS of ventilator-Associated lower respiratory tract infections (MIMOSA) Study Group. Association Between Type of Immunosuppression and the Incidence, Microbiology, and Outcomes of Bacterial Ventilator-Associated Lower Respiratory Tract Infections: A Retrospective Multicenter Study. Crit Care Med. 2025 May 1;53(5):e1080-e1094. doi: 10.1097/CCM.0000000000006615. Epub 2025 Feb 21. PMID 39982132
- [Derived] Rouze A, Lemaitre E, Martin-Loeches I, Povoa P, Diaz E, Nyga R, Torres A, Metzelard M, Du Cheyron D, Lambiotte F, Tamion F, Labruyere M, Boulle Geronimi C, Luyt CE, Nyunga M, Pouly O, Thille AW, Megarbane B, Saade A, Magira E, Llitjos JF, Ioannidou I, Pierre A, Reignier J, Garot D, Kreitmann L, Baudel JL, Voiriot G, Plantefeve G, Morawiec E, Asfar P, Boyer A, Mekontso-Dessap A, Makris D, Vinsonneau C, Floch PE, Marois C, Ceccato A, Artigas A, Gaudet A, Nora D, Cornu M, Duhamel A, Labreuche J, Nseir S; coVAPid study group. Invasive pulmonary aspergillosis among intubated patients with SARS-CoV-2 or influenza pneumonia: a European multicenter comparative cohort study. Crit Care. 2022 Jan 4;26(1):11. doi: 10.1186/s13054-021-03874-1. PMID 34983611
- [Derived] Rouze A, Martin-Loeches I, Povoa P, Metzelard M, Du Cheyron D, Lambiotte F, Tamion F, Labruyere M, Boulle Geronimi C, Nieszkowska A, Nyunga M, Pouly O, Thille AW, Megarbane B, Saade A, Diaz E, Magira E, Llitjos JF, Cilloniz C, Ioannidou I, Pierre A, Reignier J, Garot D, Kreitmann L, Baudel JL, Fartoukh M, Plantefeve G, Beurton A, Asfar P, Boyer A, Mekontso-Dessap A, Makris D, Vinsonneau C, Floch PE, Weiss N, Ceccato A, Artigas A, Bouchereau M, Duhamel A, Labreuche J, Nseir S; coVAPid Study Group. Early Bacterial Identification among Intubated Patients with COVID-19 or Influenza Pneumonia: A European Multicenter Comparative Clinical Trial. Am J Respir Crit Care Med. 2021 Sep 1;204(5):546-556. doi: 10.1164/rccm.202101-0030OC. PMID 34038699
- [Derived] Nseir S, Martin-Loeches I, Povoa P, Metzelard M, Du Cheyron D, Lambiotte F, Tamion F, Labruyere M, Makris D, Boulle Geronimi C, Pinetonde Chambrun M, Nyunga M, Pouly O, Megarbane B, Saade A, Goma G, Magira E, Llitjos JF, Torres A, Ioannidou I, Pierre A, Coelho L, Reignier J, Garot D, Kreitmann L, Baudel JL, Voiriot G, Contou D, Beurton A, Asfar P, Boyer A, Thille AW, Mekontso-Dessap A, Tsolaki V, Vinsonneau C, Floch PE, Le Guennec L, Ceccato A, Artigas A, Bouchereau M, Labreuche J, Duhamel A, Rouze A; coVAPid study group. Relationship between ventilator-associated pneumonia and mortality in COVID-19 patients: a planned ancillary analysis of the coVAPid cohort. Crit Care. 2021 May 25;25(1):177. doi: 10.1186/s13054-021-03588-4. PMID 34034777